CLINICAL TRIAL: NCT06587685
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study to Assess the Efficacy and Safety of PG-011 Gel With 8 Weeks Treatment and Extension Safety Study to 52 Weeks in Adolescents and Adults With Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of PG-011 Gel in Adolescents and Adults With Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prime Gene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG-011-AD-301; CTR20230499 (Other: http://www.chinadrugtrials.org.cn/index.html)
Record Dates: First submitted 2024-08-14; First posted 2024-09-19 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; PG-011; Pumecitinib; Atopic; Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PG-011Gel 3% (Experimental): Topically administered Pumecitinib Gel 3% to the skin twice daily for 52 or 44 weeks
  Interventions: Drug: PG-011Gel
- Vehicle Gel (Placebo Comparator): Topically administered the Vehicle Gel to the skin twice daily for 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PG-011Gel — Twice daily for 52 weeks or 44 weeks
  Other Names: PG-011Gel 3%
  Arms: PG-011Gel 3%
Drug: Vehicle — Vehicle Gel twice daily for 8 weeks
  Other Names: placebo
  Arms: Vehicle Gel

SUMMARY:
This is a Multicenter, Randomized, Double-blind, Placebo-controlled seamless and adaptive-designed phase IIb/III study to Assess the Efficacy and Safety of topical use of PG-011 Gel in adolescents and Adults With Atopic Dermatitis. It consists of phase IIb and phase III parts, phase IIb is a dose-ranging part and has been done, and phase III is a pivotal study part which is registered this time.

The goal of this phase III clinical trial is to learn if PG-011gel works to treat mild to moderate Atopic Dermatitis in adolescents and adults by topical use. It will also learn about the safety of PG-011gel. Investigators will compare PG-011gel to a placebo (a look-alike substance that contains no drug) to see if PG-011gel works to treat mild to moderate Atopic Dermatitis.

Participants will:

* Use PG-011gel or a placebo twice daily for initial 8 weeks, and followed by using PG-011 gel for all of the participants till 52-week.
* Visit the clinic at weeks 1, 2, 4 and 8 for checkups and tests, and followed by visiting the clinic every 4 weeks till 52-week.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter clinical trial in adolescent and adult participants aged from 12 to 75 years old (including threshold) with mild to moderate Atopic Dermatitis. Approximately 472 participants will be randomized 3:1 to PG-011 gel 3% BID, or placebo gel. In addition, approximately 10% of the overall study population will consist of adolescents. Participants with AD involvement of 3% to 20% BSA and IGA score of 2 to 3 will receive blinded study treatment for 8 weeks followed by an open-label treatment for 44 weeks, at last the safety follow-up for 2 weeks.

The study is to evaluate the efficacy and long-term safety of PG-011 gel 3% in the treatment of mild to moderate Atopic Dermatitis and the PK characteristics by sparse sampling.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years old≤ age ≤ 75 years old (including threshold), male or female.
2. Participants diagnosed of atopic dermatitis (AD) as defined by the Williams diagnostic criteria.
3. AD/eczema duration of at least 1 year for adults and 6 months for adolescents.
4. IGA score of 2 (mild) or 3 (moderate) at the screening day and day 1.
5. %BSA (excluding the scalp) with AD involvement of at least 10% and up to 20%.
6. Willingness to avoid pregnancy or fathering children based on the criteria as outlined in the protocol.

Exclusion Criteria:

1. Participant has unstable course of AD (spontaneously improving or rapidly deteriorating).
2. Immunocompromised (e.g. lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome).
3. Any other concomitant skin disorder(e.g. generalized erythroderma, Netherton syndrome, acne, psoriasis, urticaria, pigmentation or extensive scarring）, in the opinion of investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
4. Participant with chronic or acute infection needs to be treated with systemic antibiotics, antiviral drugs, antiparasitic drugs, anti-antigenic animal drugs or antifungal drugs within 2 weeks before randomization.
5. Participant with active acute/chronic bacterial, fungal or viral skin infections (such as herpes simplex, herpes zoster, chickenpox, etc.) before randomization, including but not limited to clinically significant secondary infections of AD or other infections associated with AD lesions.
6. Participant has human immunodeficiency virus (HIV) infection, active hepatitis C virus (HCV) infection (anti-HCV positive), active hepatitis B virus (HBV) infection (HBV-DNA > 2000IU/ml) or Treponema pallidum antibody positive and showing active.
7. Clinically significant or uncontrolled cardiovascular disease (including but not limited to unstable angina, acute myocardial infarction, heart failure, arrhythmia requiring treatment or uncontrolled hypertension).
8. Participant has serious diseases or complications of the central nervous system, respiratory system, liver, kidney, gastrointestinal tract, urinary system, endocrine system or immune system, blood system, etc., and in the opinion of the investigator, may affect the judgment of efficacy and safety .
9. Participant has mental illness such as anxiety disorder, depression, or other conditions that affect the compliance and may interfere with the implementation of clinical research.
10. Participant has a history of malignant tumors before randomization.
11. Participant has severe and uncontrolled disease that may affect safety, trial compliance, affect the evaluation of endpoints, and require the use of drugs that are not allowed in the protocol.
12. Female participant who is lactating or pregnant at the time of screening.
13. Any situation affects the safety and efficacy evaluation of the study drug judged by investigator.
14. Any other condition that, in the opinion of the investigator or sponsor, makes the subject unsuitable for participation in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieved Eczema Area and Severity Index (EASI 75) at Week 8 | 8-week
  Defined as ≥ 75% improvement in Eczema Area and Severity Index score. The EASI score ranges from 0 to 72, higher score indicates greater severity.

SECONDARY OUTCOMES:
Key Secondary Outcome: Investigators Global Assessment (IGA) score of 0/1 at Week 8 | 8-week
  Proportion of participants achieving Investigators Global Assessment (IGA) score of clear (0) or almost clear (1) with at least a 2-point decrease from baseline at Week 8.
Proportion change of eczema area and severity index (EASI) at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Proportion change in the eczema area and severity index (EASI) total score from baseline at each scheduled visit. The EASI score ranges from 0 to 72, higher score indicates greater severity.
Change of eczema area and severity index (EASI) score at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Value change in the eczema area and severity index (EASI) total score from baseline at each scheduled visit. The EASI score ranges from 0 to 72, higher score indicates greater severity.
Change from baseline of Itch Numeric Rating Scale (NRS) at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The Itch NRS is an assessment tool that participants used to report the intensity of their itch during a 24-hour recall period. The NRS score ranges from 0 to 10 points, higher score indicates greater intensity.
Proportion change from baseline of Child Dermatology Life Quality Index (CDLQI) score at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Child Dermatology Life Quality Index (CDLQI) are designed to measure the impact of any skin disease on the lives of children. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity.
Change from baseline of Child Dermatology Life Quality Index (CDLQI) score at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Child Dermatology Life Quality Index (CDLQI) are designed to measure the impact of any skin disease on the lives of children. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity.
Change from baseline of the Patient-oriented eczama Measure (POEM) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The Patient-oriented eczama Measure (POEM) is a comprehensive assessment of the patient own assessment of clinical symptoms in the past week. The POEM score ranges from 0 to 28 points, higher score indicate greater severity.
Proportion change from baseline of affected body surface area (BSA) at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Total body surface area(BSA) is 100%, and the proportion of affected body surface area(BSA) is ranged from 0 to100%, higher value indicates greater severity.
Proportion change from baseline of the Patient-oriented Eczama Measure (POEM) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The Patient-oriented Eczama Measure (POEM) is a comprehensive assessment of the patient own assessment of clinical symptoms in the past week. The POEM score ranges from 0 to 28 points, higher score indicate greater severity.
Proportion change from baseline in Scoring Atopic Dermatitis (SCORAD) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Scoring Atopic Dermatitis(SCORAD) is a tool to assess the extent and severity of eczema and will be completed before, during, and after treatment has begun to determine whether the treatment has been effective. The SCORAD score ranges from 0 to 103, and higher score indicates greater severity.
Change from baseline in Scoring Atopic Dermatitis (SCORAD) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Scoring Atopic Dermatitis(SCORAD) is a tool to assess the extent and severity of eczema and will be completed before, during, and after treatment has begun to determine whether the treatment has been effective. The SCORAD score ranges from 0 to 103, and higher score indicates greater severity.
Change from baseline of Dermatology Life Quality Index (DLQI) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Dermatology Life Quality Index (DLQI) is designed to measure the impact of any skin disease on the lives of adults.The DLQI score ranges from 0 to 30 points, higher score indicates greater severity.
Proportion change from baseline of Dermatology Life Quality Index (DLQI) score at each scheduled visit. | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Dermatology Life Quality Index (DLQI) is designed to measure the impact of any skin disease on the lives of adults.The DLQI score ranges from 0 to 30 points, higher score indicates greater severity.
The average time of the sites achieving Investigators Global Assessment(IGA) 0/1 from baseline | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Average time to achieve Investigators Global Assessment (IGA) score of clear (0) or almost clear (1) by using PG-011gel or a placebo. The IGA score ranges from 0 to 4 points, higher score indicates greater severity.
The average time of the sites achieving Investigators Global Assessment (IGA) 0/1 with at least a 2-point decrease from baseline | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Average time to achieve Investigators Global Assessment (IGA) score of clear (0) or almost clear (1) with at least a 2-point decrease from baseline by using PG-011gel or a placebo. The IGA score ranges from 0 to 4 points, higher score indicates greater severity.
Proportion of achieving Investigators Global Assessment (IGA) 0/1 at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The IGA score ranges from 0 to 4 points, higher score indicates greater severity.
Proportion of achieving Investigators Global Assessment (IGA) 0/1 with at least a 2-point decrease from baseline at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The IGA score ranges from 0 to 4 points, higher score indicates greater severity.
The average time of achieving Investigators Global Assessment (IGA) 0/1 at the atopic dermatitis (AD) target site | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The target site is a representative site of atopic dermatitis skin lesions selected by the investigator. The Investigators Global Assessment (IGA) score ranges from 0 to 4 points, higher score indicates greater severity. The IGA score 0 means clear and IGA score 1 means almost clear.
The average time of achieving Investigators Global Assessment (IGA) 0/1 with at least a 2-point decrease from baseline at the atopic dermatitis (AD) target site | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The target site is a representative site of atopic dermatitis skin lesions selected by the investigator. The Investigators Global Assessment (IGA) score ranges from 0 to 4 points, higher score indicates greater severity. The IGA score 0 means clear and IGA score 1 means almost clear.
Proportion of participants achieving at least a 3-point decrease of Itch Numeric Rating Scale (NRS) from baseline at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The Itch NRS is an assessment tool that participants used to report the intensity of their itch during a 24-hour recall period. The Itch Numeric Rating Scale(NRS) score ranges from 0 to 10 points, higher score indicates greater intensity.
Proportion of participants achieving at least a 4-point decrease of Itch Numeric Rating Scale (NRS) from baseline at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The Itch NRS is an assessment tool that participants used to report the intensity of their itch during a 24-hour recall period. The Itch Numeric Rating Scale(NRS) score ranges from 0 to 10 points, higher score indicates greater intensity.
Change from baseline of affected Body Surface Area (BSA) at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  Total Body Surface Area(BSA) is 100%, and the proportion of affected BSA is ranged from 0 to100%, higher value indicates greater severity.
Proportion of achieving Investigators Global Assessment (IGA) 0/1 in Atopic Dermatitis (AD) target site at each scheduled visit | Week1,2,4,8,12,16,20,24,28,32,36,40,44,48 and 52
  The target site is a representative site of atopic dermatitis skin lesions selected by the investigator. The Investigators Global Assessment (IGA) score ranges from 0 to 4 points, higher score indicates greater severity. The IGA score 0 means clear and IGA score 1 means almost clear.
Proportion of Investigators Global Assessment (IGA) 0/1 with at least a 2-point decrease from baseline in Atopic Dermatitis (AD) target site at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The target site is a representative site of atopic dermatitis skin lesions selected by the investigator. The Investigators Global Assessment (IGA) score ranges from 0 to 4 points, higher score indicates greater severity. The IGA score 0 means clear and IGA score 1 means almost clear.
Proportion of participants achieving Eczema Area and Severity Index(EASI) 50 at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Defined as at least 50% improvement from baseline in Eczema Area and Severity Index(EASI) score at each scheduled visit.The EASI score ranges from 0 to 72, higher score indicates greater severity.
Proportion of participants achieving Eczema Area and Severity Index(EASI) 75 at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Defined as at least 75% improvement from baseline in Eczema Area and Severity Index(EASI) score at each scheduled visit. The EASI score ranges from 0 to 72, higher score indicates greater severity.
Proportion of participants achieving Eczema Area and Severity Index(EASI) 90 at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Defined as at least 90% improvement from baseline in Eczema Area and Severity Index(EASI) score at each scheduled visit.The EASI score ranges from 0 to 72, higher score indicates greater severity.
Proportion of participants achieving Eczema Area and Severity Index(EASI) 100 at each scheduled visit | Week 1, 2,4, 8, 12,16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Defined as at least 100% improvement from baseline in Eczema Area and Severity Index(EASI) score at each scheduled visit.The EASI score ranges from 0 to 72, higher score indicates greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Study Chair — First Hospital of China Medical University; ZhiQiang Xie, Professor, Principal Investigator — Beijing Hospital; Litao Zhang, Principal Investigator — Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital; Yunsheng Liang, Principal Investigator — Dermatology Hospital of Southern Medical University; Wenli Feng, Principal Investigator — Second Hospital of Shanxi Medical University; Chao Ji, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Aie Xu, Principal Investigator — Hangzhou Third People's Hospital; Bingjiang Lin, Principal Investigator — First Affiliated Hospital of Ningbo University; Lei Cao, Principal Investigator — Brief Introduction of Wuxi No.2 People's Hospital; Rixin Chen, Principal Investigator — NANYANG FIRST PEOPLE'S HOSPITAL NATIONAL THIRD CLASS A HOSPITAL; Liming Wu, Principal Investigator — Affiliated Hangzhou First People's Hospital， School of Medicine，WestLake University; Yanyan Fen, Principal Investigator — Chengdu Second People's Hospital; Yingxia He, Principal Investigator — GENERTEC LIAOYOUGEM FLOWER HOSPITAL; Guoqiang Zhang, Principal Investigator — The First Hospital of Hebei Medical University; Meiying Jiang, Principal Investigator — Second Affiliated Hospital of Nanchang University; Linfeng Li, Principal Investigator — Beijing Friendship Hospital; Wenli Yang, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Zudong Meng, Principal Investigator — Shiyan Renmin Hospital; Kunpeng Bian, Principal Investigator — Nanyang Central Hospital
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IGA, Investigator's Global Assessment — https://www.eczemacouncil.org/investigator-global-assessment-scale.